CLINICAL TRIAL: NCT06569160
Title: Impact du déploiement de Dispositifs d'Inactivation Des pathogènes de l'Air Par UVGI Dans la Lutte Contre Les Maladies Respiratoires Touchant Les résidents d'EHPAD
Brief Title: Efficacy of Ultraviolet Germicidal Irradiation Devices to Reduce Respiratory Infections in Nursing Homes: Cluster Randomized Crossover Trial
Acronym: RESPROTECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Emile Roux (Other)
Collaborators: ANRS | French National Research Agency on Emerging Infectious Diseases (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RIPH2_GADEA_RESPROTECT
Record Dates: First submitted 2024-07-25; First posted 2024-08-23 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Infections
Keywords: Ultraviolet Germicidal Irradiation (UVGI); respiratory infections; nursing homes; elderly; cluster randomized crossover trial
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UVGI Active during period 1, UVGI Sham during period 2 (Other)
  Interventions: Device: Upper-room UVGI (Ultra-Violet Germicidal Irradiation)
- UVGI Sham during period 1, UVGI Active during period 2 (Other)
  Interventions: Device: Upper-room UVGI (Ultra-Violet Germicidal Irradiation)

INTERVENTIONS:
Device: Upper-room UVGI (Ultra-Violet Germicidal Irradiation) — Nursing homes are equipped with UVGI devices in all common living places. UVGI devices can be deactivated by installing an invisible internal filter. The inactivation filters will be installed by a technical team independent of the investigation team. Inactivation will therefore be carried out blind to the care givers and the investigation team. The centers included will be randomized into two arms. In arm A: the UVGI device will be left active during period 1, and filtered/deactivated during period 2. In arm B: the UVGI device will be filtered/deactivated during period 1 and left active during period 2.
  The two periods will last 7 months each, and will take place two years in a row on the same dates (October 1 to April 30). They will be separated by a 5-month wash-out period (May 1 to September 30), during which all UVGI equipments will be switched off in both arms.

SUMMARY:
RESPROTECT is a trial aimed at evaluating the effectiveness of upper room ultraviolet devices in reducing the frequency of severe respiratory infections in elderly nursing homes. The study takes place in 12 nursing homes in the center of France. It started in October 2024, and its final results will be availble by mid-2026.

DETAILED DESCRIPTION:
The objective of this clinical trial is to determine whether ultraviolet germicidal irradiation (UVGI) can decrease the frequency of severe acute respiratory infections in elderly people living in nursing homes.

12 elderly nursing homes (ENH) will participate in the study. In all the ENHs included, UVGI devices will be installed in upper part under the ceiling of common rooms (refectories, group activity rooms, lounges) at the start of the study. The UVGI devices can be deactivated by installing an invisible internal filter. The inactivation filters will be installed by a technical team independent of the investigation team. Inactivation will therefore be carried out blind to the care givers and the investigation team.

The nursing homes included will be randomized into two arms:

* In arm A: the UVGI device will be left active during period 1, and filtered/deactivated during period 2.
* In arm B: the UVGI device will be filtered/deactivated during period 1 and left active during period 2.

The two periods will last 7 months each, and will take place two years in a row on the same dates (October 1 to April 30). They will be separated by a 5-month wash-out period (May 1 to September 30), during which all UVGI devices will be switched off in both arms.

The main questions the study aims to answer is: do active UVGI devices decrease the number of acute respiratory infections leading to oxygen therapy, hospitalization or death during the study periods.

ELIGIBILITY:
Center Inclusion criteria:

Elderly Nursing homes (ENH):

* Having a system for monitoring cases of upper and lower respiratory infections among their residents.
* Agreeing to take part in the study
* Undertaking to comply with the protocol
* Accepting the installation of UVGI devices
* Undertaking to provide all residents or their legal guardians/curators with an individual information leaflet.

Center Exclusion criteria:

ENH:

* Not wishing to be equipped with UVGI devices in all rooms considered necessary to be equipped by the investigators
* Having planned a major change to the structure (extension, renovation, closure, requalification, etc.) during the course of the study, which could affect the study population and/or UVGI air treatment devices.

Individual Inclusion criteria:

All residents present in one of the participating ENH at the start of each of the two study periods, or arriving in one of the participating ENH during one of the two periods, will be eligible

Individual Exclusion criteria :

Residents of the ENH included in the study who have expressed (personally or through a relative or legal representative) the wish that their personal data not be used for the study will not be included in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe acute symptomatic upper and lower respiratory infections | From enrollment to the end of the second follow-up period (19 months later)
  Acute symptomatic upper and lower respiratory infections include: sinusitis, otitis media, nasopharyngitis, angina, tracheitis, bronchitis, pneumonia, pulmonary abscesses and COPD exacerbations. Symptomatic infection with SARS-Cov-2 will be considered by default as a respiratory infection, even if extra-respiratory symptoms predominate.
  Severe acute respiratory infections = acute respiratory infections leading to oxygen therapy, hospitalization or death.

SECONDARY OUTCOMES:
Incidence of acute upper and lower respiratory infections, all grades of severity combined | From enrollment to the end of the second follow-up period (19 months later)
  Acute symptomatic upper and lower respiratory infections include: sinusitis, otitis media, nasopharyngitis, angina, tracheitis, bronchitis, pneumonia, pulmonary abscesses and COPD exacerbations. Symptomatic infection with SARS-Cov-2 will be considered by default as a respiratory infection, even if extra-respiratory symptoms predominate.
Incidence of all-cause hospitalisations or death | From enrollment to the end of the second follow-up period (19 months later)
  All-cause hospitalisations or death include hospitalisation due to acute respiratory infections, hospitalisations due to any other documented or undocumented cause, death to acute respiratory infections, and deaths from any other documented or undocumented cause
Viral and bacterial load in air samples | From enrollment to the end of the second follow-up period (19 months later)
  Air samples collected every 7 weeks in 2 common living areas per center
Viral and bacterial load on fomites samples | From enrollment to the end of the second follow-up period (19 months later)
  Samples collected every 7 weeks in 2 common living areas per center
Incremental Cost-effectiveness ratio | From enrollment to the end of the second follow-up period (19 months later)
  Generated/avoided costs
Incidence of adverse events of interest, overall and by severity grade | From enrollment to the end of the second follow-up period (19 months later)
  Adverse events of interest: keratitis and erythematous skin eruptions in body areas exposed to light

CONTACTS AND LOCATIONS:
Overall Officials: Cyril CORNILLE, MD, Principal Investigator — Hôpital Emile Roux, le Puy en Velay
Locations (12):
- France (12):
  - EHPAD Notre Dame, Beaulieu
  - EHPAD du Centre hospitalier du Pays de Craponne sur Arzon, Craponne-sur-Arzon
  - EHPAD Paradis, Espaly-Saint-Marcel
  - EHPAD du Centre hospitalier Pierre Gallice, Langeac
  - EHPAD Les Terrasses de la Gazeille, Le Monastier-sur-Gazeille
  - EHPAD Les Patios du Velay, Le Puy-en-Velay
  - EHPAD Nazareth, Le Puy-en-Velay
  - EHPAD Saint-Joseph, Le Puy-en-Velay
  - EHPAD L'Age d'Or, Monistrol-sur-Loire
  - EHPAD Résidence Sigolène, Sainte-Sigolène
  - EHPAD Saint Jacques, Saugues
  - EHPAD Marie Goy, Vorey

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study protocol, SAP and ICF: start date 1st July 2025. No end date. CSR: start date 1st July 2026. No end date.
  IPD: 1st October 2026. No end date.
Access Criteria: Study protocol, SAP and ICF: free access on clinicaltrials.gov IPD: on demand to trial team. Approval by the Scientific Advisory Board.

DOCUMENTS (2):
  • Study Protocol (2025-09-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT06569160/Prot_002.pdf
  • Statistical Analysis Plan (2025-09-30): https://cdn.clinicaltrials.gov/large-docs/60/NCT06569160/SAP_003.pdf